CLINICAL TRIAL: NCT04269083
Title: A Biomarker-driven Therapeutic Strategy for Esophageal Cancer, the BoRgES Trial: a Multicenter Randomized Phase II Study of BIRC3-expression Directed Preoperative Chemoradiotherapy in Patients With Resectable Adenocarcinoma of the ESophagus and Esophagogastric Junction
Brief Title: A Biomarker-driven Therapeutic Strategy for Esophageal Cancer Chemoradiotherapy in Patients With Resectable Adenocarcinoma of the ESophagus and Esophagogastric Junction
Acronym: BoRgES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GR-2016-02361134
Record Dates: First submitted 2020-02-06; First posted 2020-02-13 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-02

CONDITIONS: Esophageal Cancer
Keywords: esophageal-gastric junction cancer, preoperative chemoradiotherapy, BIRC3
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: open-label, multicenter, randomized phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): fresh specimens from the tumour and normal mucosa will be collected endoscopically at diagnosis and placed immediately into RNALater to isolate RNA. The mRNA expression of BIRC3 will be quantified using a SYBR green-based real-time PCR analysis; the BIRC3 median expression in normal mucosa samples will be used as calibrator. Patients with a tumor expression level of BIRC3 lower than the established cutoff will receive a standard carboplatin/paclitaxel regimen with concurrent radiotherapy followed by surgery. Patients with an expression of BIRC3 higher or equal than the cutoff (chemoradiation resistant patients) will undergo upfront surgery.
  Interventions: Other: BIRC3
- control arm (Active Comparator): fresh specimens from the tumour and normal mucosa will be collected endoscopically at diagnosis and placed immediately into RNALater to isolate RNA. The mRNA expression of BIRC3 will be quantified using a SYBR green-based real-time PCR analysis; the BIRC3 median expression in normal mucosa samples will be used as calibrator. Patients with a tumor expression level of BIRC3 lower than the established cutoff will receive a standard carboplatin/paclitaxel regimen with concurrent radiotherapy followed by surgery. Patients with an expression of BIRC3 higher or equal than the cutoff (chemoradiation resistant patients) will undergo upfront surgery.
  Interventions: Other: BIRC3

INTERVENTIONS:
Other: BIRC3 — BIRC3-expression directed preoperative chemoradiotherapy in patients with resectable adenocarcinoma of the esophagus and EGJ

SUMMARY:
Preoperative chemoradiotherapy followed by surgery has been accepted as the standard of care for resectable adenocarcinoma of the esophagus and esophagogastric junction (EGJ). However, in a large part of the cases the tumor is extremely resistant to chemoradiotherapy, and those patients do not benefit from this treatment but are exposed to its negative consequences such as toxicity and delayed surgical therapy. The hypothesis is that a biomarker-driven therapeutic strategy in which patients will receive preoperative chemoradiotherapy or upfront surgery based on the basal tumor expression of BIRC3 could improve the R0 resection rate if compared with a standard strategy in unselected patients.

DETAILED DESCRIPTION:
BoRgES trial is a multicenter, randomized phase II study of BIRC3-expression directed preoperative chemoradiotherapy in patients with resectable adenocarcinoma of the esophagus and EGJ. The main objective of this proposal is to provide evidence for a novel therapeutic strategy with enormous significance for patients affected by this disease.

Only a part of the patients with esophageal adenocarcinoma benefit from neoadjuvant therapy, and the clinical efficacy of chemoradiotherapy is reduced by the pre-existence of cellular drug resistance. Thus, there is an urgent need to identify patients who could not benefit from preoperative treatment. The study will define an innovative therapeutic strategy directed by the expression of BIRC3 as a predictive marker for discriminating patients who will most likely be resistant to preoperative chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the esophagus and EGJ (Siewert I/II) surgical resectable (cT2-4a, N0-1, M0), as determined by Endoscopic Ultra Sound (EUS) and or PET-TC scan. cT1N1 tumors are eligible, T1N0 tumors and in situ carcinoma are not eligible.
* If tumor extends below the EGJ junction into the proximal stomach, the bulk of the tumor must involve the esophagus or GE junction. The tumor must not extend more than 2 cm into the stomach (Siewert III). Gastric cancers with minor involvement of the GE junction or esophagus are not eligible.
* Age >18, no age upper limit unless patient would be unable to tolerate chemoradiotherapy.
* Have given written informed consent prior to any study-specific procedures.
* ECOG performance status 0-2.
* No prior thoracic radiotherapy allowed.
* Adequate hematological, renal, cardiac, hepatic and pulmonary functions.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-05-24 (Estimated); Primary Completion 2024-03-24 (Estimated); Study Completion 2024-08-24 (Estimated)

PRIMARY OUTCOMES:
R0, number of patients achieving R0 resection. | 3 years
  number of patients achieving R0 resection.

SECONDARY OUTCOMES:
OS | 3 years
  overall survival
DFS | 3 years
  disease free survival
tumour response | 3 years
  tumour response evaluated either by Mandard's tumour regression grade
safety profile | 3 years
  safety profile (incidence of ≥ grade 3 adverse events using Common Terminology Criteria for Adverse Events - CTCAE - version 4.0).

IPD SHARING:
Plan to Share IPD: No